CLINICAL TRIAL: NCT00095329
Title: A Phase I/II, Open-Label Pilot Trial to Evaluate the Safety of Rapamune (Sirolimus) in Patients With Multiple Sclerosis
Brief Title: Treating Multiple Sclerosis With Sirolimus, an Immune System Suppressor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT AMS02
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: relapsing-remitting MS; nonresponsive to standard of care MS; sirolimus
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sirolimus (Experimental)
  Interventions: Biological: sirolimus

INTERVENTIONS:
Biological: sirolimus

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the drug sirolimus in patients with multiple sclerosis (MS) who have failed other treatments.

DETAILED DESCRIPTION:
MS is a chronic autoimmune disease of the central nervous system in which myelin, the protein sheath that protects nerve cells, is degraded by T cells and macrophages, leading to an eventual loss of neurologic function. MS can be classified as either relapsing-remitting, in which patients experience worsening in symptoms followed by partial or complete recovery of function; or progressive, in which patients have a gradual increase in symptoms, with or without relapses. Standard treatments used to treat relapsing-remitting MS are only modestly effective and may be associated with significant toxicity. There is a need to develop therapies with lower toxicities that can be administered early during the course of disease and have the potential to stop disease progression altogether. Sirolimus has been demonstrated to provide potent immunosuppression in recent clinical trials involving kidney transplantation, and may help people with autoimmune diseases like MS. This study will determine the benefit of sirolimus in MS patients.

Blood and urine collection will occur at screening. Participants will take daily doses of sirolimus for 6 months. There will be nine study visits; they will occur at Days 14, 28, 42, 56, 90, 120, 150, 180, and 225. Medication adverse events, concomitant medications, and vital signs will be recorded at Visits 1 through 8. At all visits, patient compliance to the sirolimus regimen will be measured, and blood and urine collection will occur. Physical and neurological exams, magnetic resonance imaging (MRI) brain scans, MS status tests, and a chest x-ray will be conducted at selected times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS
* Evidence of demyelination on magnetic resonance imaging (MRI) scan
* Expanded Disability Status Scale (EDSS) score between 0 and 6
* Nonresponsive to beta-interferon or Glatiramer acetate therapy
* Discontinuation of beta-interferon or Glatiramer acetate therapy within 1 month prior to study entry
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Primary progressive MS
* Prior treatment with immunosuppressants
* Steroid therapy within 1 month prior to study entry
* Evidence of active infection or cancer
* Heart or hematologic dysfunction
* High levels of lipids in the blood
* Use of lipid-lowering agents
* History of cirrhosis or liver disease requiring treatment
* History of hepatitis B or C
* Active cytomegalovirus infection
* Kidney disease requiring treatment
* Active lung disease
* Diabetes
* Hyperthyroidism
* HIV infection
* Tuberculosis
* History of alcohol or drug abuse within 6 months prior to study entry
* Claustrophobia or inability to undergo MRI
* Pregnancy or breast-feeding

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Safety of sirolimus, including number of lesions detected by brain MRI
Tolerability of sirolimus
Mean number of new and overall total number of gadolinium-enhancing lesions reported on sequential brain MRIs

SECONDARY OUTCOMES:
Efficacy, as measured by change in the mean number of new and overall total number of gadolinium-enhancing lesions on pre-treatment brain MRIs, compared to post-treatment
Effect of sirolimus therapy on the immune function of patients with relapsing-remitting multiple sclerosis (RRMS)

CONTACTS AND LOCATIONS:
Overall Officials: Samia J. Khoury, MD, Principal Investigator — Center for Neurological Diseases, Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Center for Neurological Diseases, Brigham and Women's Hospital, Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Background] Meier DS, Weiner HL, Khoury SJ, Guttmann CR. Magnetic resonance imaging surrogates of multiple sclerosis pathology and their relationship to central nervous system atrophy. J Neuroimaging. 2004 Jul;14(3 Suppl):46S-53S. doi: 10.1177/1051228404266268. PMID 15228759
- [Background] Gonsette RE. New immunosuppressants with potential implication in multiple sclerosis. J Neurol Sci. 2004 Aug 15;223(1):87-93. doi: 10.1016/j.jns.2004.04.025. PMID 15261567
- [Background] Lucchinetti C, Bruck W. The pathology of primary progressive multiple sclerosis. Mult Scler. 2004 Jun;10 Suppl 1:S23-30. doi: 10.1191/1352458504ms1027oa. PMID 15218806
- [Background] Kovarik JM, Burtin P. Immunosuppressants in advanced clinical development for organ transplantation and selected autoimmune diseases. Expert Opin Emerg Drugs. 2003 May;8(1):47-62. doi: 10.1517/14728214.8.1.47. PMID 14610911
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/